CLINICAL TRIAL: NCT01728766
Title: Longitudinal Studies of Breast Milk Zinc Transfer to Appropriate- and Small-for-gestational-age, Predominantly Breast Fed, Bangladeshi Infants
Brief Title: Breast Milk Zinc Transfer to Appropriate- and Small-for-gestational-age Bangladeshi Infants
Status: Completed | Type: Observational
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-035
Record Dates: First submitted 2012-11-04; First posted 2012-11-20 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2012-11

CONDITIONS: Small for Gestational Age at Delivery; Post-term Infant, Not Heavy-for-dates
Keywords: Breast milk zinc transfer; Bangladeshi infants; appropriate-for-gestational-age; small-for-gestational-age; plasma zinc

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Breast milk Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants under-6 months and their mothers: Small for gestational age at delivery. Post-term Infant, Not Heavy-for-dates.
  Interventions: Other: Small for gestational age at delivery; Other: Post-term Infant, Not Heavy-for-dates

INTERVENTIONS:
Other: Small for gestational age at delivery — Small for gestational age at delivery. gestational age at >37 weeks by and birth weight <2500 g
  Other Names: Small-for-Gestational Age (SGA)
Other: Post-term Infant, Not Heavy-for-dates — Appropriate for gestational age at delivery. Gestational age at >37 weeks and birth weight >2800 g
  Other Names: Appropriate-for-gestational age (AGA)

SUMMARY:
Data collected from this study will provide information on the breast milk zinc concentration, maternal and infant zinc status, and transfer of zinc from mothers breast milk to infants during first six months of life.

DETAILED DESCRIPTION:
The International Atomic Energy Agency (IAEA) has reviewed published literature to collect information for its Coordinated Research Project (CRP) on Zinc Nutrition During Early Life , and observed that there is limited information on: 1) the concentration of zinc in breast milk of mothers in lower income countries at different times post-partum; 2) the total amount of zinc transferred from mothers to infants at different ages in these settings, and 3) zinc transfer from mother to infant born with appropriate-for-gestational-age (AGA) and small-for-gestational-age (SGA). Therefore, IAEA has planned to assist local scientists to collect such information from selected countries. The International Zinc Nutrition Consultative Group (IZiNCG) has identified Bangladesh as a country with high risk of zinc deficiency (IZiNCG, 2004), where the rate of SGA infants is >30% - one of the highest in the world (de Onis, 1998). Thus, Bangladesh is an appropriate candidate country to participate in this CRP.

This study will enroll 50 healthy, full-term, newborn infants (>37 weeks gestational age by ultrasound) and their mothers if they plan to breast-feed exclusively for at least 4 months and also to continue breast feeding for at least 12 months. The infants will be examined, weighed and measured within 48 hours of birth, half of whom will be AGA (BW>2800g) and the other half SGA (BW<2500g). Infants with any acute or chronic illnesses, or congenital anomalies will not be eligible. Any mother with toxaemia, pregnancy-induced hypertension, multiple pregnancies, previously diagnosed as positive for HIV/hepatitis B infections, or habituated to smoking or alcohol consumption will also be excluded. The participants will be recruited from Nandipara, Dhaka, an urban community where the ICDDRB has ongoing clinical study facilities.

Each of the eligible mother-infant pairs will be studied in 3 separate rounds, at 4, 12 and 24 weeks post-partum. In each round, two-week studies of breast milk transfer from the mother to the infant will be carried out, using the deuterium "dose-to-the-mother" technique. In each round, the women will be requested to attend the Dhaka Hospital of ICDDR, B on day 0, for collection of baseline saliva samples from mother-infant pairs and administration of deuterium to the mothers. Study health workers will make home visits on days 1, 2, 3, 4, 13, and 14 and collect saliva samples from the infants and their mothers on days 1, 2, 13 and 14, of each round.

~2 ml of saliva will be collected for each sample from both the mother and the infant.

On days 0 and 4 of each round, 5-10 ml of manually-expressed breast milk will be collected for determining their zinc concentration. The total zinc transfer from mother to infant will be calculated as the product of the mean daily milk volume, as determined from the deuterium studies, and the mean milk zinc concentration on the days of milk collection.

On the first day of each of the rounds at 4, 12 and 24 week post-partum 2.0 ml of venous blood will be collected from both the mothers and infants for serum zinc assay.

Body weight, length and head circumference of infants, and body weight and height of mothers will be measured on day 0 at 4, 12 and 24 week post-partum.

Breast milk volume and zinc concentration, and total zinc transfer from mothers to infants will be the major outcome variables, which will be examined for conformance to the normal distribution and transformed if required. Means of the major outcome variables will be compared for AGA and SGA infants for each time points, using repeated measures ANOVA. Repeated measures analysis of covariance will be used to assess if these relationships change with age. Analyses will be done with SAS Release 9 and SPSS version 10.

ELIGIBILITY:
Inclusion Criteria:

* AGA, birth weight >2800 g at ≥37 weeks of gestation
* SGA, birth weight <2500 g at ≥37 weeks of gestation

Exclusion Criteria:

* Other than the above birth weight
* Any congenital anomalies abnormalities, chronic infections as were infants with c, or acute illnesses at the time of enrollment
* Mothers with pregnancy-induced hypertension, multiple pregnancies, known HIV or hepatitis B infection, or use of tobacco products or alcohol were excluded from the study,

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants were 46 mothers and their term infants, 20 of whom were classified as appropriate for gestational age (AGA, birth weight >2800 g at ≥37 weeks of gestation) and 26 of whom were classified as small for gestational age (SGA, birth weight <2500 g at ≥37 weeks of gestation). Gestational age was assessed by ultrasonography at ~32 weeks of gestation. Only mothers who were planning to breast feed exclusively for at least four months were included in the study. Mothers with pregnancy-induced hypertension, multiple pregnancies, known HIV or hepatitis B infection, or use of tobacco products or alcohol were excluded from the study, as were infants with congenital abnormalities, chronic infections, or acute illnesses at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Amount of zinc transferred through breast milk | at 4, 12 and 24 weeks after delivery of the infants
  During each round of study, a milk sample was collected during the visit to icddr,b on study day 1 and 5. On each occasion, the breast was cleansed with soap and water and rinsed with copious amounts of deionized water. The milk sample was then collected ~2-3 minutes after the feeding was initiated by momentarily removing the infant from the breast, so the study assistant could manually express 5-10 mL milk into a zinc-free beaker. The milk sample was then transferred to a plastic screw cap vial and transported to the laboratory, as described above for the saliva samples. The milk zinc concentration was measured by atomic absorption spectrometer (AAS, AA6501S, Shimadzu, Kyoto, Japan). The total zinc transfer from mother to infant was calculated as the product of the mean daily milk volume, as determined from the deuterium tracer studies, and the mean milk zinc concentration on the corresponding milk collection days.

SECONDARY OUTCOMES:
Plasma zinc content of both the mother and the infant | at 4, 12 and 24 weeks after the delivery of the infants
  On the first morning of each round, 2 mL of venous blood was drawn from both the mother and infant for plasma zinc analyses, using stainless steel needles and certified trace element-free, evacuated collection tubes (Sarstedt LiH monovette, Sarstedt, Newton, NC, USA). The infant samples were drawn 90 minutes after the first morning feeding, but the mothers' samples were not timed in relation to meals. The plasma was separated within 60 minutes and stored at -20o C until analysis. The plasma samples were diluted (1:12) with distilled, deionized water, vortexed, and analyzed using the same AAS described above. The plasma samples were also compared with commercially available standard zinc nitrate solution (BDH, England), bi-level control serum (Cat # 66816; UTAK Laboratories Inc, Valencia, CA), and pooled serum to determine the accuracy and precision of the analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Dr M Munirul Islam, MBBS, PhD, Principal Investigator — Associate Scientist
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh ( icddr,b),, Dhaka, Bangladesh

REFERENCES:
- [Derived] Islam MM, Brown KH. Zinc transferred through breast milk does not differ between appropriate- and small-for-gestational-age, predominantly breast-fed Bangladeshi infants. J Nutr. 2014 May;144(5):771-6. doi: 10.3945/jn.113.189308. Epub 2014 Mar 5. PMID 24598881